CLINICAL TRIAL: NCT05598021
Title: Instrumental Evaluation of Self-correction in Patients With Juvenile and Adolescent
Brief Title: Self-correction Evaluation in Scoliosis Patients
Status: Recruiting | Type: Observational
Sponsor: Istituto Scientifico Italiano Colonna Vertebrale (Other)
Responsible Party: Sponsor
Other Study IDs: Self-correction
Record Dates: First submitted 2022-10-21; First posted 2022-10-28 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Scoliosis; Juvenile; Scoliosis; Adolescence
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ultrasound assessment: Quantitative comparison between ultrasound images performed in active self-correction and in a spontaneous position
- RX assessment: Quantitative comparison between radiological images performed in active self-correction and in a spontaneous position

SUMMARY:
To date, there is no objective assessment method for the quality of the self-correction performed by patients with scoliosis.

The study consists of two parts, both retrospective, and distinct on the basis of the tools used to assess self-correction.

Part 1: Retrospective assessment of the radiographic variations between spontaneous position and self-correction in subjects suffering from juvenile and adolescent idiopathic scoliosis. Both measurements were performed in a single session.

Part 2: Retrospective assessment of the variations between spontaneous and self-correcting position in subjects with juvenile and adolescent idiopathic scoliosis using objective parameters deriving from non-invasive 3D ultrasound instrumentation (Scolioscan, Telefeld, Hong Kong).

ELIGIBILITY:
Inclusion Criteria for both parts:

* Diagnosis of juvenile or adolescent idiopathic scoliosis;
* Age >= 10 years;
* Single and double curves with amplitude >= 15 ° Cobb;
* Performing exercises according to SEAS for at least 6 months

Only for part 1 (radiographic)

* Availability of radiographic investigation in upright position and in self-correction Only for part 2 (ultrasound)
* Availability of ultrasound assessment in upright position and in self-correction
* Complete radiograph of the spine in anteroposterior projection performed in the 45 days preceding or following the medical examination.
* Risser between 0 and 2.

Exclusion Criteria:

For both parts:

* Patients with more than 2 scoliotic curves
* Patients with secondary scoliosis
* Patients suffering from learning disabilities or clinical conditions impairing neuromotor control
* Patients lacking the necessary measures to evaluate the outcome.

Part 2 only (ultrasound)

● Patients undergoing brace treatment

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with adolescent and juvenile idiopathic scoliosis.
Sampling Method: Non-Probability Sample
Enrollment: 185 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Self-correction measure | through study completion, an average of 6 months
  The angular difference of the curves resulting from the detection with Scolioscan or Rx in the spontaneous position compared to what was obtained in the same condition but in the self-correcting position.

CONTACTS AND LOCATIONS:
Locations (1):
- ISICO, Milan, Mi, Italy

IPD SHARING:
Plan to Share IPD: Undecided